CLINICAL TRIAL: NCT05044546
Title: Pilot Study to Evaluate a Behavioral Activation Prenatal and Postpartum Intervention for Depressed Pregnant Smokers
Brief Title: A Behavioral Activation Prenatal and Postpartum Intervention for Depressed Pregnant Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0972; NCI-2021-07469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0972 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); R01DA014301 (NIH); R01MH076776 (NIH); R01MH087692 (NIH); R34DA048265 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2021-09-14 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Depression; Tobacco Use Disorder
MeSH Terms: conditions — Depression; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Aim 1 and secondary aim 2 (focus group) (Experimental): Participants participate in focus group over 60-90 minutes. Participants who completed and dropped out of postpartum treatment also participate in a focus group.
  Interventions: Procedure: Discussion
- Aim 3 Group I (BA) (Experimental): Participants participate in smoking cessation counseling over 15 minutes and BA counseling sessions over 45 minutes once a week for 10 weeks to pilot test delivery via smart phone videoconferencing and to conduct process evaluation of technical issues in use of smart phones.
  Interventions: Behavioral: Behavioral Activation Therapy; Other: Tobacco Cessation Counseling
- Aim 3 Group II (HW) (Experimental): Participants participate in smoking cessation counseling over 15 minutes and health and wellness education counseling sessions over 45 minutes once a week for 10 weeks to pilot test delivery via smart phone videoconferencing and to conduct process evaluation of technical issues in use of smart phones.
  Interventions: Behavioral: Health Education; Other: Tobacco Cessation Counseling
- Aim 4 Group III (BA) (Experimental): During the prenatal period, participants of 18-22 weeks gestational age will receive 10 individual sessions with 15 minutes of smoking cessation counseling ad 45 minutes of behavioral activation counseling sessions. These women will have 16 weeks to complete their 10 individual sessions.
  Interventions: Behavioral: Behavioral Activation Therapy; Other: Questionnaire Administration; Other: Tobacco Cessation Counseling
- Aim 4 Group IV (HW) (Experimental): During the prenatal period, participants of 18-22 weeks gestational age will receive 10 individual sessions with 15 minutes of smoking cessation counseling and 45 minutes of health and wellness education counseling sessions. These women will have 16 weeks to complete their 10 individual sessions.
  Interventions: Behavioral: Health Education; Other: Questionnaire Administration; Other: Tobacco Cessation Counseling

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy — Participate in BA counseling
  Other Names: BAT; Behavioral Activation
  Arms: Aim 3 Group I (BA); Aim 4 Group III (BA)
Procedure: Discussion — Participate in focus group
  Other Names: Discuss
  Arms: Aim 1 and secondary aim 2 (focus group)
Behavioral: Health Education — Participate in health and wellness education counseling
  Arms: Aim 3 Group II (HW); Aim 4 Group IV (HW)
Other: Questionnaire Administration — Ancillary studies
  Arms: Aim 4 Group III (BA); Aim 4 Group IV (HW)
Other: Tobacco Cessation Counseling — Participate in smoking cessation counseling
  Arms: Aim 3 Group I (BA); Aim 3 Group II (HW); Aim 4 Group III (BA); Aim 4 Group IV (HW)

SUMMARY:
This study evaluates a mood management and health and wellness smoking cessation intervention for depressed pregnant smokers during and after birth. This study may help pregnant smokers who are experiencing depression quit smoking and stay smoke-free after their babies are born.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct qualitative group interviews with depressed pregnant smokers and depressed smokers within the first 4 months of the postpartum period, to adapt and refine the delivery of behavioral activation therapy (BA) and health and wellness education (HW) via smart phone videoconferencing, a BA and HW smart phone application (app) including supportive smoking cessation messages in the prenatal and postpartum periods. (Stage IA) II. Adapt BA and smoking cessation counseling manuals, BA and HW app and content, and treatment integrity rating scales for the prenatal and postpartum period. (Stage IA) III. Pilot test the delivery, via smart phone videoconferencing, of a 10-week treatment course of BA and HW and conduct process evaluation of technical issues in the use of smart phones, barriers to participation and retention; completion of study assessments, and; adequacy of procedures for addressing psychiatric emergencies. (Stage IA)

III. Conduct a preliminary randomized trial with depressed pregnant smokers comparing BA to HW to evaluate:

IIIa. Effect of BA on abstinence at 4 1/2 months postpartum. (Stage IB) IIIb. Effect of BA on depression at 4 1/2 months postpartum. (Stage IB) IIIc. Feasibility of acceptance of the smart phone delivery of BA and HW, and assessment components indicated by a) retention; b) completion of prenatal and postpartum sessions; c) completion of study assessments, d) strength of therapeutic alliance from both the participant and therapist perspective; e) participant and therapist ratings on satisfaction questionnaire. (Stage IB) IIId. Feasibility of study procedures as indicated by a) percentage of sessions interrupted by technical difficulties, and; b) percentage of urine cotinine tests and/or anabasine tests received for biochemical verification of self-reported abstinence at 4 1/2 months postpartum. (Stage IB)

SECONDARY OBJECTIVES:

I. Evaluate change in hypothesized treatment mechanisms including positive affect, negative affect, and cognitive function in relation to treatment effects on smoking and depression. (Stage IB) II. Conduct qualitative interviews with women who completed and did not complete postpartum treatment to assess a) barriers to completing treatment sessions; b) usefulness of postpartum treatment; c) suggestions for decreasing barriers and improving treatment acceptability, and; d) relevant experiences unexpected by participants and researchers. (Stage IB)

OUTLINE:

AIM 1 AND SECONDARY AIM 2: Participants participate in focus group over 60-90 minutes. Participants who completed and dropped out of postpartum treatment also participate in a focus group.

AIM 3: Participants are assigned to 1 of 2 groups.

GROUP I (BA): Participants participate in smoking cessation counseling over 15 minutes and BA counseling sessions over 45 minutes once a week for 10 weeks to pilot test delivery via smart phone videoconferencing and to conduct process evaluation of technical issues in use of smart phones.

GROUP II (HW): Participants participate in smoking cessation counseling over 15 minutes and health and wellness education counseling sessions over 45 minutes once a week for 10 weeks to pilot test delivery via smart phone videoconferencing and to conduct process evaluation of technical issues in use of smart phones.

AIM 4: Participants are randomized to 1 of 2 groups.

GROUP III (BA): During the prenatal period, participants of 18-22 weeks gestational age will receive 10 individual sessions with 15 minutes of smoking cessation counseling ad 45 minutes of behavioral activation counseling sessions. These women will have 16 weeks to complete their 10 individual sessions.

During the prenatal period, participants of 23-32 weeks gestational age will receive 10 individual sessions with 15 minutes of smoking cessation counseling and 45 minutes of behavioral activation counseling sessions. These women will have 12 weeks to complete their 10 individual sessions.

We may do additional check in calls or text communications with participants to maintain engagement between prenatal and postpartum treatment sessions.

Following birth, women may have up to a month break before resuming individual sessions, though have the option to resume earlier if preferred. Women will receive an additional 4counseling sessions in postpartum over 6 weeks. The participants will complete 1 follow up visit that occurs 4 ½ months postpartum.

GROUP IV (HW): During the prenatal period, participants of 18-22 weeks gestational age will receive 10 individual sessions with 15 minutes of smoking cessation counseling and 45 minutes of health and wellness education counseling sessions. These women will have 16 weeks to complete their 10 individual sessions.

During the prenatal period, participants of 23-32 weeks gestational age will receive 10 individual sessions with 15 minutes of smoking cessation counseling and 45 minutes of health and wellness education counseling sessions. These women will have 12 weeks to complete their 10 individual sessions.

We may do additional check in calls or text communications with participants to maintain engagement between prenatal and postpartum treatment sessions.

Following birth, women may have up to a month break before resuming individual sessions, though have the option to resume earlier if preferred. Women will receive an additional 4counseling sessions in postpartum over 6 weeks. The participants will complete 1 follow up visit that occurs 4 ½ months postpartum.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Aim 1

1. Pregnant (or within 4 months post-partum for aim 1 only)
2. Meets criteria for current Major Depressive Disorder (MDD) as assessed by the Mini International Neuropsychiatric Interview (MINI) 7.0.2 OR PHQ score of 10 or greater.
3. ≥ 18 years of age
4. Have a telephone
5. Self report smoking, even a puff, cigarettes, little cigars and/or Cigarillos in the past 30 days.
6. Approximately two thirds of the sample will be gestational age up to 36 weeks, and approximately one third will be within 4 months postpartum
7. Able to speak and read English
8. Subjects must report a current residence in the State of Texas

Eligibility Criteria: AIM 3 Inclusion criteria for Aims 3

1. Meets criteria for current Major Depressive Disorder (MDD) as assessed by the Mini International Neuropsychiatric Interview (MINI) 7.0.2 OR PHQ score of 10 or greater.
2. ≥ 18 years of age
3. Have an address and telephone number where they may be reached
4. Self report smoking, even a puff, cigarettes, little cigars and/or Cigarillos in the past 30 days.
5. Gestational age between 12 to 34 weeks
6. Able to speak and follow verbal and written instructions in English
7. Subjects must report a current residence in the State of Texas and must not have plans to move out of the state in the next 2.5 months
8. Subjects referred directly from UT Health providers, the provider or designee will confirm pregnancy status through their electronic health record prior to the referral. Subjects referred by any other means will confirm positive pregnancy status through an at-home test.
9. Willing to refrain from the use of other nicotine/tobacco products for the duration of the study
10. Agree to be treated via telehealth (live audio-video conference and phone) and to be contacted via text and/or email
11. Provide informed consent and agree to all assessments and study procedures

Exclusion Criteria:

Exclusion criteria for Aims 1

1. Rated on the Columbia-Suicide Severity Rating Scale113 at screening as in the past month having had active suicidal ideation with some intent to act or active suicidal ideation with specific plan and intent (indicated by answering "YES" on both Q3 and Q4, and/or 5) and/or endorsing "YES" to having engaged in preparatory acts towards or attempting suicide in the past 3 months (as indicated by answering "YES" to both parts of Q6)
2. Have a lifetime or current diagnosis of Psychotic Disorder as assessed by specified Mini International Neuropsychiatric Interview (MINI) 7.0.2 modules.
3. Have a past or current diagnosis of Bipolar Disorder I or II or have a past or current diagnosis of Other specified Bipolar and related disorder as assessed by specified MINI 7.0.2 modules.
4. Any otherwise not specified medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
5. Participant considered by the investigator as unsuitable candidate for full participation in the study.

Exclusion criteria for Aim 3

1. Currently participating in individual psychotherapy
2. Currently participating in other smoking cessation treatments and refuses to refrain from use for the duration of the study
3. Rated on the Columbia-Suicide Severity Rating Scale113 at screening as in the past month having had active suicidal ideation with some intent to act or active suicidal ideation with specific plan and intent (indicated by answering "YES" on both Q3 and Q4, and/or 5) and/or endorsing "YES" to having engaged in preparatory acts towards or attempting suicide in the past 3 months (as indicated by answering "YES" to both parts of Q6)
4. Have a lifetime or current diagnosis of Psychotic Disorder as assessed by specified Mini International Neuropsychiatric Interview (MINI) 7.0.2 modules.
5. Have a past or current diagnosis of Bipolar Disorder I or II or have a past or current diagnosis of Other specified Bipolar and related disorder as assessed by specified MINI 7.0.2 modules.
6. Any otherwise not specified medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
7. Participant considered by the investigator as unsuitable candidate for full participation in the study.

Eligibility Criteria: AIM 4 Inclusion criteria for AIM 4

1. Meets criteria for current Major Depressive Disorder (MDD) as assessed by the Mini International Neuropsychiatric Interview (MINI) 7.0.2 OR PHQ score of 10 or greater.
2. ≥ 18 years of age
3. Have an address and telephone number where they may be reached
4. Self report smoking, even a puff, cigarettes, little cigars and/or Cigarillos in the past 30 days.
5. Gestational age between 18to 32 weeks
6. Able to speak and follow verbal and written instructions in English
7. Subjects must report a current residence in the State of Texas and must not have plans to move out of the state in the next 7-8 months
8. Subjects will confirm positive pregnancy status through study provided pregnancy test or provide paperwork verifying pregnancy status if the pregnancy test is inconclusive
9. Willing to refrain from the use of other nicotine/tobacco products for the duration of the study
10. Agree to be treated via telehealth (live audio-video conference and phone) and to be contacted via text and/or email
11. Provide informed consent and agree to all assessments and study procedures
12. Interested in treatment that might change smoking behavior or help them quit smoking
13. Be the only participant in their household currently receiving treatment on this protocol

Exclusion criteria for Aim 4

1. Currently participating in individual psychotherapy
2. Currently participating in other smoking cessation treatments and refuses to refrain from use for the duration of the study
3. Rated on the Columbia-Suicide Severity Rating Scale113 at screening as in the past month having had active suicidal ideation with some intent to act or active suicidal ideation with specific plan and intent (indicated by answering "YES" on both Q3 and Q4, and/or 5) and/or endorsing "YES" to having engaged in preparatory acts towards or attempting suicide in the past 3 months (as indicated by answering "YES" to both parts of Q6)
4. Have a lifetime or current diagnosis of Psychotic Disorder as assessed by specified Mini International Neuropsychiatric Interview (MINI) 7.0.2 modules.
5. Have a past or current diagnosis of Bipolar Disorder I or II or have a past or current diagnosis of Other specified Bipolar and related disorder as assessed by specified MINI 7.0.2 modules.
6. Any otherwise not specified medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
7. Participant considered by the investigator as unsuitable candidate for full participation in the study.

Inclusion criterion for Secondary Aim 2, Stage IB Women enrolled in the study who dropped out of the study during the first month of the postpartum treatment phase or women who completed at least 3 of the 4 postpartum treatment sessions Because study therapists will be asked to complete the WAI and acceptability of treatment ratings as part of Aim 4 work, they will be considered study participants and will provide verbal consent to complete these measures.

Inclusion criterion for Study Therapists

1. Masters degree in psychology, social work, or other counseling degree
2. Training in the delivery of psychotherapy and counseling interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2027-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Minnix, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AIM 1: Qualitative Focus Groups/Individual Interviews: Qualitative group/individual interviews to refine delivery of BA and HW therapy conditions via smartphone
- Aim 3: Assigned HW Control: 10 week treatment course of Health and Wellness Educational Therapy (Control Condition) delivered via smartphone videoconferencing
- Aim 3: Assigned BA Treatment: 10 week treatment course of Behavioral Activation therapy (Treatment Condition) delivered via smartphone videoconferencing
- Aim 4: Health and Wellness (HW): Standard smoking cessation counseling plus HW, a didactic health education counseling on ways women can physically care for themselves during pregnancy and postpartum.
- Aim 4: Behavioral Activation (BA): Standard smoking cessation counseling plus BA, which focuses on increasing rewarding and adaptive behaviors and decreasing avoidance and withdrawal.
Period: Aim 1
Arm/Group | AIM 1: Qualitative Focus Groups/Individual Interviews | Aim 3: Assigned HW Control | Aim 3: Assigned BA Treatment | Aim 4: Health and Wellness (HW) | Aim 4: Behavioral Activation (BA)
Started | 11 | 0 | 0 | 0 | 0
Completed | 11 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: AIM 3 Pilot Study
Arm/Group | AIM 1: Qualitative Focus Groups/Individual Interviews | Aim 3: Assigned HW Control | Aim 3: Assigned BA Treatment | Aim 4: Health and Wellness (HW) | Aim 4: Behavioral Activation (BA)
Started | 0 | 3 | 6 | 0 | 0
Completed | 0 | 3 | 5 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Period: AIM 4: Randomized Trial
Arm/Group | AIM 1: Qualitative Focus Groups/Individual Interviews | Aim 3: Assigned HW Control | Aim 3: Assigned BA Treatment | Aim 4: Health and Wellness (HW) | Aim 4: Behavioral Activation (BA)
Started | 0 | 0 | 0 | 3 | 3
Completed | 0 | 0 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AIM 1: Focus Groups: Qualitative group/individual interviews to refine delivery of BA and HW therapy conditions via smartphone
- AIM 3: Women Assigned to Health & Wellness (HW): 10 week treatment course of Health and Wellness Educational Therapy (Control Condition) delivered via smartphone videoconferencing
- AIM 3: Women Assigned to Behavioral Activation (BA): 10 week treatment course of Behavioral Activation Treatment Condition delivered via smartphone videoconferencing
- AIM 4: Health & Wellness (HW); AIM 4: Behavioral Activation (BA): Standard smoking cessation counseling plus HW, a didactic health education counseling on ways women can physically care for themselves during pregnancy and postpartum.
- Total: Total of all reporting groups
Arm/Group | AIM 1: Focus Groups | AIM 3: Women Assigned to Health & Wellness (HW) | AIM 3: Women Assigned to Behavioral Activation (BA) | AIM 4: Health & Wellness (HW) | AIM 4: Behavioral Activation (BA) | Total
Number analyzed (Participants) | 11 | 3 | 6 | 3 | 3 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 6 | 3 | 3 | 26
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 6 | 3 | 3 | 26
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 10 | 3 | 5 | 2 | 2 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 1 | 3 | 1 | 1 | 14
  White | 2 | 2 | 1 | 2 | 1 | 8
  More than one race | 0 | 0 | 2 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 3 | 6 | 3 | 3 | 26

OUTCOME MEASURES:

1. Primary Outcome: Abstinence
Description: Point-prevalence abstinence at last treatment visit at 10 weeks or earlier if ppt was lost to follow up defined as both a self-report of not smoking during the previous 7 days and a negative result from biochemical verification.
Time Frame: Last treatment visit at 10 weeks or earlier if participant was lost to follow up
Population: Analysis was not a part of AIM 1.
Measure: Count of Participants; unit: Participants
Groups:
- AIM 3: Assigned Health & Wellness (HW): Standard smoking cessation counseling plus HW, a didactic health education counseling on ways women can physically care for themselves during pregnancy and postpartum.
- Aim 3: Assigned Behavioral Activation: Standard smoking cessation counseling plus BA, which focuses on increasing rewarding and adaptive behaviors and decreasing avoidance and withdrawal
Arm/Group | AIM 3: Assigned Health & Wellness (HW) | Aim 3: Assigned Behavioral Activation
Number analyzed (Participants) | 3 | 6
Participants | 2 | 1

2. Primary Outcome: Depression
Description: Depression as assessed using the Patient Health Questionnaire (PHQ-9) measure. The PHQ 9 is the major depressive episode scale from the Patient Health Questionnaire (PHQ). There are nine items on the Patient Health Questionnaire (PHQ-9). The PHQ-9 Depression Severity score is calculated by assigning score of 0, 1, 2, 3 to the response category of "not at all", "several days", "more than half, the days", and "nearly every day", respectively. The PHQ-9 total score for the nine items ranges from 0 to 27. The higher the value indicates a more severe score. The total score is a combination of the number of total symptoms experienced and the frequency of those symptoms over a two week period. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe, and severe depression, respectively. There are no subscales on the PHQ-9
Time Frame: Last treatment visit at 10 weeks or eariler if participant was lost to follow up
Population: Analysis was not a part of AIM 1.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | AIM 3: Assigned Health & Wellness (HW) | Aim 3: Assigned Behavioral Activation
Number analyzed (Participants) | 3 | 6
Scores on a Scale | 2 (1.41) | 7 (3.54)

3. Primary Outcome: Abstinence
Description: Point-prevalence abstinence at 4 ½ months postpartum follow-ups defined as both a self-report of not smoking during the previous 7 days and a negative result from biochemical verification.
Time Frame: 4 ½ months postpartum
Population: Analysis was not a part of AIM 1 & AIM 3 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | AIM 4: Health & Wellness (HW) | AIM 4: Behavioral Activation (BA)
Number analyzed (Participants) | 3 | 3
Participants | 2 | 1

4. Primary Outcome: Depression
Description: as for outcome 2
Time Frame: 4 1/2 months postpartum
Population: Analysis was not a part of AIM 1 & AIM 3 for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIM 4: Health & Wellness (HW) | AIM 4: Behavioral Activation (BA)
Number analyzed (Participants) | 3 | 3
scores on a scale | 0.67 (1.15) | 7.34 (10.21)

ADVERSE EVENTS:
Time Frame: Adverse event monitoring will stop at the final treatment visit, or earlier if the ppt withdraws or becomes lost to follow up. AIM 3, AEs were collected for an average of 11 months. For AIM 4, AEs were collected for an average of 7.5 months.
Description: Only psychiatric adverse events, whether or not related to the treatment, will be reported. AIM 1 was qualitative data, therefore no adverse events were collected.
Arm/Group | AIM 3: Women Assigned to Health & Wellness (HW) | AIM 3: Women Assigned to Behavioral Activation (BA) | AIM 4: Health & Wellness (HW) | AIM 4: Behavioral Activation (BA)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT05044546/Prot_SAP_000.pdf